CLINICAL TRIAL: NCT02915055
Title: Multimodal Analgesia With NSAID vs. Narcotics Alone for Post-operative Meniscectomy: A Prospective Observational Study
Brief Title: NSAID vs. Narcotics
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-01645
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Multimodal Analgesia; Nonsteroidal Anti-inflammatory Drugs
Keywords: Analgesic efficacy; knee arthroplasty; Opioid consumption; Pain Medicine; Narcotics; Multimodal Analgesia
MeSH Terms: interventions — Ibuprofen; Acetaminophen; oxycodone-acetaminophen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pain following knee arthroscopic meniscectomy
  Interventions: Drug: Ibuprofen 600 mg; Drug: standard oxycodone/acetaminophen

INTERVENTIONS:
Drug: Ibuprofen 600 mg — Ibuprofen 600 mg to be taken every 8 hours (TID) as needed (PRN
Drug: standard oxycodone/acetaminophen
  Other Names: Percocet

SUMMARY:
This will be a single-center, prospective observational study. The study will compare post-operative pain scores and narcotic consumption between two groups of patients - one cohort will receive ibuprofen (Motrin) and Percocet (to be used as needed) while the other cohort will receive only Percocet. Both pain management options are considered to be standard of care.

The primary objective of the study is to compare patients' reported pain and narcotic use following meniscectomy, and determine if NSAIDs can provide adequate pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* ASA class I-II
* Patients scheduled for meniscectomy

Exclusion Criteria:

* Contraindication to ibuprofen or oxycodone/acetaminophen (e.g. hypersensitivity, history of GI or bleeding disorder)
* Legally incompetent or mentally impaired (e.g. minors, Alzheimer's subjects, dementia, etc.)
* Younger than 18 years of age or older than 65
* Any patient considered a vulnerable subject
* Patients on pain medication prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients indicated for isolated arthroscopic meniscectomy will be identified from the operating room schedules of orthopaedic surgeons participating in the study. And a review of patients' medications and past medical histories will be performed based on their electronic medical records to identify any current pain medications or exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) score | 4 Hours
  Scale consisting of a drawn line from 0 to 100 - you will be asked to mark where you believe your pain is (100 being worse pain).
Pain Verbal Rating Scale | 4 Hours
  Verbal rating scale, consisting of 4 points (0 = no pain, 1 = mild, 2 = moderate, and 3 = severe).

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Campbell, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States